CLINICAL TRIAL: NCT00303758
Title: Essai Randomise Comparant Deux Stategies De Chimiotherapie Dans Les Cancers Pancreatiques Avances: LV5FU2 Simplifie + Cisplatine Suivi de Gemcitabine, Versus Gemcitabine Suivi de LV5FU2 Simplifie + Cisplatine en Can de Progression
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic Pancreatic Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000453841; FFCD-0301; EU-20543
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2006-12

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cisplatin; Fluorouracil; Gemcitabine; Leucovorin

ARMS (2):
- LV5FU2 simplifié + cisplatine puis gemcitabine si progression (Active Comparator): LV5FU2 simplifié + cisplatine puis gemcitabine si progression
  Interventions: Drug: cisplatin; Drug: fluorouracil; Drug: gemcitabine hydrochloride; Drug: leucovorin calcium
- gemcitabine puis LV5FU2 simplifié + cisplatine si progression (Experimental): gemcitabine puis LV5FU2 simplifié + cisplatine si progression
  Interventions: Drug: cisplatin; Drug: fluorouracil; Drug: gemcitabine hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, leucovorin, cisplatin, and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) and giving them in different ways may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective in treating metastatic pancreatic cancer.

PURPOSE: This randomized phase III trial is studying two different combination chemotherapy regimens to compare how well they work in treating patients with metastatic pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with unresectable metastatic pancreatic cancer treated with fluorouracil, leucovorin calcium, and cisplatin followed by gemcitabine hydrochloride vs gemcitabine hydrochloride followed by fluorouracil, leucovorin calcium, and cisplatin.

Secondary

* Compare progression-free survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Compare the percentage of these patients needing second-line therapy.
* Compare the duration of hospitalization of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to ECOG performance status (0 or 1 vs 2), participating center, location of the tumor (ampullar region vs other locations), and infusion rate of gemcitabine hydrochloride (30 vs 100 minutes). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive leucovorin calcium IV over 2 hours on day 1, cisplatin IV over 1 hour on day 1 or 2, and fluorouracil IV over 46 hours on day 1 and 2. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients with disease progression also receive gemcitabine hydrochloride IV over 30 or 100 minutes weekly for 7 weeks. Patients then receive gemcitabine hydrochloride IV on days 1, 8, and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine hydrochloride IV over 30 or 100 minutes weekly for 7 weeks in the absence of disease progression or unacceptable toxicity. Patients with disease progression receive fluorouracil, leucovorin calcium, and cisplatin as in arm I.

Quality of life is assessed at baseline and then every 2 months.

After completion of study therapy, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 202 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas or ampulla

  * Metastatic disease
  * Unresectable disease
* Measurable disease, meeting the following criteria:

  * No prior radiotherapy to the only site of measurable disease
  * Diameter > 10 mm by spiral CT scan or MRI OR > 20 mm by conventional methods
* No brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 2 months
* No contraindication to chemotherapy
* Creatinine clearance > 60 mL/min
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Alkaline phosphatase < 5 times normal
* Bilirubin ≤ 3 mg/dL
* No coronary insufficiency
* No symptomatic cardiac disease
* Good hydration possible
* No Child-Pugh class B or C cirrhosis
* No other malignancy except for basal cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior palliative or adjuvant chemotherapy
* At least 4 weeks since prior radiotherapy
* No radiotherapy during or for 4 weeks after study therapy
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2005-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2012

SECONDARY OUTCOMES:
Progression-free survival | 2012
Toxicity | 2012
Quality of life | 2012
Percentage of patients needing second-line therapy | 2012
Duration of hospitalization | 2012

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Seitz, MD, Study Chair — CHU de la Timone; Jean-Louis Legoux, MD, Study Chair — Hopital Haut Leveque; Pascal Hammel, MD, PhD, Study Chair — Hopital Beaujon
Locations (46):
- France (46):
  - Centre Hospitalier d'Abbeville, Abbeville
  - Hopital Duffaut, Avignon
  - Centre Hospitalier de Blois, Blois
  - Centre Hospitalier Universitaire Ambroise Pare - Boulogne, Boulogne
  - Centre Hospitalier Docteur Duchenne, Boulogne-sur-Mer
  - C.H. Bourg En Bresse, Bourg-en-Bresse
  - Centre Hospitalier Pierre Oudot, Bourgoin
  - Centre Hospitalier Universitaire d'Amiens, Caen
  - Centre Hospitalier de Chalons-en-Champagne, Châlons-en-Champagne
  - CHR Clermont Ferrand, Hotel dieu, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Hopital Louis Pasteur, Colmar
  - Hopital Du Bocage, Dijon
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Hospitalier Draguignan, Draguignan
  - Centre Hospitalier De Dunkerque - CHD, Dunkirk
  - Centre Hospitalier Intercommunal St. Aubin les Elbeuf, Elbeuf
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Clinique Pasteur, Guilherand-Granges
  - Hopital Robert Boulin, Libourne
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Centre Hospitalier Regional et Universitaire de Lille, Lille
  - Hopital Edouard Herriot, Lyon
  - Hopital Saint Joseph, Marseille
  - CHU de la Timone, Marseille
  - CHU Nord, Marseille
  - Centre Hospitalier de Martigues, Martigues
  - Centre Hospitalier General de Mont de Marsan, Mont-de-Marsan
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CHR Hotel Dieu, Nantes
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Haut Leveque, Pessac
  - Clinique Ste - Marie, Pontoise
  - CHU - Robert Debre, Reims
  - Centre Eugene Marquis, Rennes
  - Hopital Charles Nicolle, Rouen
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Joliot Curie Des Docteurs Jean-Christophe Chardon Jacques Hernandez Et Laurent Gasnault, Saint-Martin-Boulogne
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
  - Centre Hospitalier de Semur en Auxois, Semur-en-Auxois
  - Centre Hospitalier de Soissons, Soissons
  - Hopital Universitaire Hautepierre, Strasbourg
  - Centre Hospitalier de Tarbes, Tarbes
  - Nouvelle Clinique Generale, Valence

REFERENCES:
- [Result] Dahan L, Bonnetain F, Ychou M, Mitry E, Gasmi M, Raoul JL, Cattan S, Phelip JM, Hammel P, Chauffert B, Michel P, Legoux JL, Rougier P, Bedenne L, Seitz JF; Federation Francophone de Cancerologie Digestive. Combination 5-fluorouracil, folinic acid and cisplatin (LV5FU2-CDDP) followed by gemcitabine or the reverse sequence in metastatic pancreatic cancer: final results of a randomised strategic phase III trial (FFCD 0301). Gut. 2010 Nov;59(11):1527-34. doi: 10.1136/gut.2010.216135. PMID 20947887